CLINICAL TRIAL: NCT05986227
Title: The Sequential Combination of FOLFOX and Toripalimab for Perioperative Immuno-oncology Therapy of HER2-negative Gastroesophageal Adenocarcinoma (Siewert I/II): a Multicenter, Open-label, Randomized Controlled, Phase 1b/2 Trial (SCORPIO/NCCES05)
Brief Title: The Sequential Combination of FOLFOX and Toripalimab for Perioperative Immuno-Oncology Therapy of HER2-negative Adenocarcinoma of the Esophagogastric Junction (Siewert I/II):
Acronym: SCORPIO
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022111621481500
Record Dates: First submitted 2023-04-30; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2022-11

CONDITIONS: Gastroesophageal Adenocarcinoma
Keywords: GEA

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FOLFOX(D1)was combined with toripalimab(D3) (Experimental)
  Interventions: Drug: toripalimab FOLFOX
- FOLFOX(D1)was combined with toripalimab(D1) (Experimental)
  Interventions: Drug: toripalimab FOLFOX
- FOLFOX(D3) was combined with toripalimab(D1) (Experimental)
  Interventions: Drug: toripalimab FOLFOX
- FOLFOX(D1) (Active Comparator)
  Interventions: Drug: toripalimab FOLFOX

INTERVENTIONS:
Drug: toripalimab FOLFOX — Toripalimab（3mg/kg, q2w, IV）oxaliplatin (85 mg/m2 IV), leucovorin (400 mg/m2 IV) and 5-FU (2400 mg/m2/day continuous IV infusion over 48 h)

SUMMARY:
The addition of immunotherapy to chemotherapy improves outcomes in patients with HER2-negative gastroesophageal adenocarcinoma (GEA), and investigators aim to explore its role in the perioperative setting. Moreover, optimizing the timing schedule of these two therapies is critical when balancing efficacy and safety. This Chinese, multicenter, open-label phase 1b/2 trial will evaluate the efficacy and toxicity of perioperative folinic acid, fluoro-uracil, oxali-platin (FOLFOX), and toripalimab (JS001, a novel PD-1 inhibitor) in combination at various schedules in the neoadjuvant setting in patients with HER2-negative resectable GEA: three cycles each in Arm A: FOLFOX (D1, q2w) followed by toripalimab (D3, 3 mg/kg, q2w); Arm B: concurrent FOLFOX (D1, q2w) combined with toripalimab (D1, 3 mg/kg, q2w); Arm C: toripalimab (D1, 3 mg/kg, q2w) followed by FOLFOX (D3, q2w); Arm D: FOLFOX (D1, q2w) alone. The primary end-point is the dose-limiting toxicity in Phase 1b and the pathological complete response rate in Phase 2; secondary end-points include major pathologic response, disease-free survival, and event-free survival.A fixed sample size of 126 patients is used in this study, with a safety run-in period (n = 6) and cohort expansion period (n = 24), a dropout rate of 5% within 12 months of follow-up. Each arm receives three cycles of FOLFOX (D1, q2w) followed by 15 cycles of toripalimab (D1, 240 mg, q3w) in the neoadjuvant setting. Pre-treatment biopsies, post-resection specimens, serial liquid biopsy, and gut microbiota samples on treatment will be collected to explore the biomarkers' predictive value on diverse schedule efficacy and safety.

DETAILED DESCRIPTION:
This Chinese, multicenter, open-label phase 1b/2 trial will evaluate the efficacy and toxicity of perioperative folinic acid, fluoro-uracil, oxali-platin (FOLFOX), and toripalimab (JS001, a novel PD-1 inhibitor) in combination at various schedules in the neoadjuvant setting in patients with HER2-negative resectable GEA: three cycles each in Arm A: FOLFOX (D1, q2w) followed by toripalimab (D3, 3 mg/kg, q2w); Arm B: concurrent FOLFOX (D1, q2w) combined with toripalimab (D1, 3 mg/kg, q2w); Arm C: toripalimab (D1, 3 mg/kg, q2w) followed by FOLFOX (D3, q2w); Arm D: FOLFOX (D1, q2w) alone. The primary end-point is the dose-limiting toxicity in Phase 1b and the pathological complete response rate in Phase 2; secondary end-points include major pathologic response, disease-free survival, and event-free survival. A fixed sample size of 126 patients is used in this study, with a safety run-in period (n = 6) and cohort expansion period (n = 24), a dropout rate of 5% within 12 months of follow-up. Each arm receives three cycles of FOLFOX (D1, q2w) followed by 15 cycles of toripalimab (D1, 240 mg, q3w) in the neoadjuvant setting. Pre-treatment biopsies, post-resection specimens, serial liquid biopsy, and gut microbiota samples on treatment will be collected to explore the biomarkers' predictive value on diverse schedule efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years;
* Male or Female;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
* Histologically or cytologically confirmed locally advanced adenocarcinoma of esophagus or gastroesophageal junction (Siewert type I/II);
* Human epidermal growth factor receptor 2 (HER2)-negative tumors;
* Clinical staging cT2-T4aNanyM0 or TanyN+M0 (UICC/AJCC 8th edition), potentially resectable disease;
* Adequate hematologic and end organ function based on laboratory results obtained within 14 days prior to initiation of study treatment;
* For women of childbearing potential: agreement to remain abstinent；no evidence of pregnancy within 72 hours before the start of study regimen;
* Must be willing and able to provide written informed consent.

Exclusion Criteria:

* Known unresectable disease，cT4b disease invading aorta or trachea;
* Known distant metastases，including supraclavicular lymph nodal disease；
* Uncontrollable pleural or pericardial effusion，or ascites requiring repeated interventions;
* Prior chemotherapy, immunotherapy, targeted therapy, thoracic radiotherapy or prior surgical resection for an esophageal tumor;
* Poor nutritional status, BMI < 18.5 Kg/m2; if symptomatic nutritional support is corrected before randomization, enrollment may continue to be considered after assessment by the principal investigator;
* History of allergy to biological drugs produced by Chinese hamster ovary cells, any component of toripalimab, tegafur, oxaliplatin or other platinum drugs;
* History of severe allergic, allergic reactions, or other hypersensitivity to chimeric or humanized antibodies or fusion proteins;
* Patients with prior malignancies are eligible if they have been disease-free for > 5 years and are deemed by their physician to be at low risk for recurrence. Patients with squamous or basal cell carcinoma of the skin, melanoma in situ, carcinoma in situ of the cervix, or carcinoma in situ of the colon or rectum that have been effectively treated are eligible, even if these conditions were diagnosed within 5 years prior to enrollment；
* History of any active autoimmune disease or autoimmune disease, including myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid syndrome-related vascular thrombosis, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, glomerulonephritis, etc.; hypothyroidism (hormone replacement therapy can be considered to be included);
* History of immunosuppressive drugs, or systemic hormones used to achieve immunosuppressive purposes (dose > 10 mg/day prednisone or equivalent dose) within 2 weeks before the first use of the study drug; in the absence of active autoimmune diseases, inhaled or local steroids are allowed and doses > 10 mg/day prednisone or equivalent doses of adrenocorticotropic hormone replacement;
* History of type 1 diabetes, whose blood glucose is controlled after treatment with a stable dose of insulin dosing regimen may be enrolled in this study;
* History of live attenuated vaccines are received within 4 weeks before the first use of the study drug;
* History of major surgery or severe trauma within 4 weeks before the first use of the study drug;
* History of eczema, psoriasis, lichen simplex chronicus, or dermatologic manifestations of vitiligo (eg, patients with psoriatic arthritis were excluded from the study) were permitted to enroll in this study if they met the following conditions: a) had rash coverage less than 10% of body surface area (BSA); b) had adequately controlled disease at baseline and required only low-potency topical steroid therapy; c) did not have an acute exacerbation of the underlying disease within the past 12 months without the need for PUVA (psoralen plus ultraviolet A radiation), methotrexate, retinoids, biologics, oral calcineurin inhibitors, high-titer, or oral steroid therapy for]；
* History of idiopathic pulmonary fibrosis, organizing pneumonia (such as bronchiolitis obliterans), drug-induced pneumonia, idiopathic pneumonia, interstitial pneumonia, or evidence of active pneumonia on screening chest CT scan;
* History of immunodeficiency, including HIV test positive, or suffering from other acquired or congenital immunodeficiency diseases, or a history of organ transplantation or allogeneic bone marrow transplantation;
* Uncontrolled cardiac clinical symptoms or diseases, including but not limited to: a) NYHA class II or higher heart failure; b) unstable angina; c) myocardial infarction within 1 year; d) clinically significant supraventricular or ventricular arrhythmia that remains poorly controlled without or after clinical intervention.
* Known hereditary or acquired bleeding and thrombophilia (such as hemophilia, coagulation dysfunction, thrombocytopenia, etc.);
* Known serious infection (CTCAE > 2) within 4 weeks before the first use of the study drug, such as severe pneumonia requiring hospitalization, bacteremia, infectious complications, etc.; baseline chest imaging showed active pulmonary inflammation, symptoms and signs of infection within 14 days before the first use of the study drug or oral or intravenous antibiotics, except for the prophylactic use of antibiotics;
* Active pulmonary tuberculosis infection detected by medical history or CT examination, or history of active pulmonary tuberculosis infection within 1 year before enrollment, or history of active pulmonary tuberculosis infection more than 1 year ago but without regular treatment;
* Active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (hepatitis C antibody positive, and HCV RNA above the lower limit of detection of the analytical method);
* Pregnant or lactating women;
* Other factors that may lead to forced halfway termination of the study as judged by the investigator, such as having other serious diseases (including mental illness) requiring concomitant treatment, alcoholism, drug abuse, family or social factors that may affect the safety or compliance of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
DLT | through study completion,an average of 1.5 years
  Phase 1b: safety of the combination regimen in different drug treatment sequences, i.e., dose-limiting toxicity (DLT).
PCR | 0.5 year
  Phase II: efficacy of different sequential combinations of drugs, i.e., postoperative pathological complete response rate (pCR).